CLINICAL TRIAL: NCT01659697
Title: Diabetes Prevention in Patients Aged 25-55 From Ethiopian Origin With Prediabetes: Evaluation of Feasibility and Efficacy of Intensive or Less Intensive Lifestyle Intervention
Brief Title: Diabetes Prevention in Prediabetic Patients
Acronym: DPEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 057/2012
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Ethnic Group; Young Adults; Prediabetes; Community Health Services
Keywords: lifestyle; diabetes prevention; BMI; physical activity
MeSH Terms: conditions — Prediabetic State; Motor Activity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intensive Lifestyle counseling
  Interventions: Behavioral: intensive lifestyle counseling
- usual lifestyle counseling
  Interventions: Behavioral: intensive lifestyle counseling

INTERVENTIONS:
Behavioral: intensive lifestyle counseling — Intensive lifestyle counseling will include a bi annual visit of the primary physician and nurse, a group intervention about use of medical resources, healthy lifestyle a one to one intervention with a dietician about diet and a one to one intervention with a physiotherapist about exercise

SUMMARY:
This study will evaluate the feasibility and efficacy of two interventions of lifestyle ( intensive and less intensive) to prevent diabetes in patients from Ethiopian origin, aged 25 to 55 years old with prediabetes living in Israel and insured by Clalit Health Services in the Central district, using resources existing in this Health Care system (HMO).

ELIGIBILITY:
Inclusion Criteria:

* prediabetes
* age 25-55
* ethiopian origin

Exclusion Criteria:

* diabetes
* age under 25 or above 55
* non ethiopian origin

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients aged 25-55 from Ethiopian origin leaving in Israel with pre diabetes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
occurence of diabetes | two years period
  Patients included in the study will have a one year lifestyle intervention ( two arms: intensive, less intensive) and will be followed for two years for the occurence of diabetes

SECONDARY OUTCOMES:
change in Body Mass index and Physical activity | two years

CONTACTS AND LOCATIONS:
Overall Officials: Joelle A Singer, M.D., Principal Investigator — Meir Medical Center; Dalia Blumenthal, M.D., Study Director — Meir Medical Center
Locations (1):
- Central district Clalit Health Services, Rishon LeZiyyon, Israel